CLINICAL TRIAL: NCT01552083
Title: A Community Pharmacist-led Intervention to Improve Screening of Sleep Apnea in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Etude SAS
Record Dates: First submitted 2012-01-27; First posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; screening; community pharmacy
MeSH Terms: conditions — Sleep Apnea Syndromes

INTERVENTIONS:
Other: screening of sleep apnea — 2 validated screening questionnaires (Berlin questionnaire, Epworth scale)

SUMMARY:
The purpose of this study is to evaluate the feasibility and the effectiveness of sleep apnea screening program for patients at risk in community pharmacies.

DETAILED DESCRIPTION:
Background: The sleep apnea syndrome (SAS) is a common disease but unknown. According to epidemiological studies, approximately 5% to 10% of the general population is living with SAS. Untreated sleep apnea has an important individual impact: it is accompanied by sleep disturbances and vigilance and frequent co-morbidities such as hypertension, diabetes or other cardiovascular diseases. Also, it has a cost to the community due to significant traffic accidents and work accidents more frequent in this population and weight for health insurance for cardiovascular diseases. However, its screening and its management remain largely insufficient. The report of the Ministry of Health in 2006 estimated that only 15% of subjects with a SAS would be diagnosed.

The Law "Hospital, Patients, Health and Territories" (HPST) in 2009 provides pharmacists with new responsibilities in the health screening, care coordination, or in therapeutic education (Article 38 of Law HPST).

Objective: In this dual context, this study aims to assess the feasibility and effectiveness of an information campaign and screening of SAS in patients at risk in the community pharmacies. The investigators analyze whether the involvement of community pharmacists in the care pathway of a patient at risk is effective, that is to say if it improves the detection rate and diagnostic the disease in this population.

Project Description: 400 patients at risk of SAS will be recruited by the participating pharmacists. Screening intervention consists in 2 validated questionnaires which evaluate SAS risk (Berlin Questionnaire, Epworth Sleepiness Scale). Pharmacist distributes also an information leaflet about SAS, and refers patient to general practitioner with questionnaires results. Patients are followed by the pharmacists for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Taking 1 or more anti-hypertension drugs
* Overweight (BMI > 25)
* Snoring
* Signed informed consent

Exclusion Criteria:

* To have a sleep apnea treatment
* Not to have a referent doctor
* To have a long-term illness
* Did not sign informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients referred by the general practitioner to sleep specialist for SAS diagnosis test | 6 months after the intervention of pharmacists.

SECONDARY OUTCOMES:
Satisfaction of patients and pharmacists | 6 months after the intervention of pharmacist
Proportion of patients with sleep apnea | 6 months after the intervention of pharmacists

CONTACTS AND LOCATIONS:
Overall Officials: Nathalise Pelletier-Fleury, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Cermes3, CNRS UMR8211 - Inserm U988, Villejuif, France